CLINICAL TRIAL: NCT01334593
Title: The Effect of Neoadjuvant Chemoradiotherapy on Exercise Capacity in Colrectal Cancer Patients
Brief Title: Assessment of Fitness After Neoadjuvant Chemoradiotherapy in Rectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Michelle Mossa (Other Government)
Responsible Party: Sponsor-Investigator, Michelle Mossa, Deputy Research and Development Director, Liverpool University Hospitals NHS Foundation Trust
Organization: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Other Study IDs: 11/H1002/12b
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rectal Cancer

SUMMARY:
Neoadjuvant chemoradiotherapy (NACRT) prior to surgery for lower gastrointestinal (colon and rectal) cancer is associated with improved survival, but also adversely affects physical fitness, potentially rendering patients unfit for major surgery or increasing the risk of adverse outcome (death and serious complications) after major surgery. The investigators aim to obtain pilot data showing that neoadjuvant chemoradiotherapy (NACRT)reduces objectively measured exercise capacity (fitness).

DETAILED DESCRIPTION:
Purpose: To evaluate the effects of chemoradiotherapy on pre-operative fitness of patients prior to major colorectal cancer surgery.

Design: Patients will act as their own case-control.

Patients will be consented at the earliest available opportunity following the decision that they have surgically treatable disease and they consent to pre-operative NACRT. Consent for the study will be gained as an outpatient. At "visit 1" patients will undergo CPET, as is our current standard practice, prior to commencing neoadjuvant chemoradiotherapy. As part of the assessment, they will have pulmonary function testing (static lung volumes, lung diffusing capacity). They will then undergo 6 weeks of long course NACRT, as is standard current practice at our institution. At "visit 2", approximately four to six weeks following chemoradiotherapy another CPET test will be repeated. This is also current standard practice at our institution. Data from visit 1 and visit 2 will be compared in a paired manner. A statistician will be consulted to assess the degree of normality of the data, the statistical tests to use, and for power calculations. At no point will any treatments be postponed or changed solely for the purposes of collecting data for the research.

ELIGIBILITY:
Inclusion Criteria:

* All patients listed to undergo neoadjuvant chemoradiotherapy for downstaging of colorectal cancer, with a view to undergo elective colorectal surgery at Aintree University Hospitals.

Exclusion Criteria:

* Unable to consent.
* Under 18 years of age.
* Significant ischaemic changes of >1.5mm symptomatic and > 2mm asymptomatic observed on routine cardiopulmonary exercise test.
* Any other absolute contraindications to CPET based on the ATS guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer is the third commonest cause of cancer related death (after breast and lung cancer) in the United Kingdom and the second commonest in non smokers. Around 100 new cases of colorectal cancer are diagnosed each day in the UK. In 2002 there were 34,889 new cases of colorectal cancer diagnosed in the United Kingdom, and approximately 17,000 deaths (CRUK 2006). Almost three quarters of bowel cancer cases occur in people aged 65 and over. Within England, mortality rates are generally higher in the north of the country.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Measurement of Cardio Pulmonary exercise test related parameters (VO2 at AT) pre and post neoadjuvant chemoradiotherapy in rectal cancer patients. | 2 years
  Exercise capacity (fitness) before and after NACRT will be assessed using CPET.We have pilot data on an upper gastrointestinal cancer cohort that shows that neoadjuvant chemotherapy alone results in lower levels of fitness (mean fall VO2@LT of 2.19ml/kg/min), which relates to survival before stomach and oesophageal surgery in a group of patients in Liverpool. These data also suggest that the insult of chemotherapy and surgery increases mortality

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm A West, Principal Investigator — Aintree University Hospitals NHS Foundation Trust, Liverpool, UK
Locations (1):
- Aintree University Hospitals, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Derived] West MA, Loughney L, Barben CP, Sripadam R, Kemp GJ, Grocott MP, Jack S. The effects of neoadjuvant chemoradiotherapy on physical fitness and morbidity in rectal cancer surgery patients. Eur J Surg Oncol. 2014 Nov;40(11):1421-8. doi: 10.1016/j.ejso.2014.03.021. Epub 2014 Apr 12. PMID 24784775